CLINICAL TRIAL: NCT07340047
Title: Clinical Trial of H1ssF Vaccine vs. Seasonal Influenza Vaccine in Previously Unvaccinated Adults and Previously Vaccinated Adults
Brief Title: H1ssF Flu Vaccine Clinical Trial
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDIM-2025-31286
Record Dates: First submitted 2025-12-09; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Influenza
Keywords: Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- H1ssF vaccine (Experimental)
  Interventions: Biological: H1ssF vaccine
- Flucelvax seasonal vaccine (Active Comparator)
  Interventions: Biological: Flucelvax seasonal vaccine

INTERVENTIONS:
Biological: H1ssF vaccine — Experimental influenza vaccine
  Arms: H1ssF vaccine
Biological: Flucelvax seasonal vaccine — Licensed influenza vaccine
  Arms: Flucelvax seasonal vaccine

SUMMARY:
This is a two-arm, open-label, randomized, phase 1, controlled clinical trial intended to evaluate the safety and immunologic response to the experimental vaccine H1ssF (H1 stabilized stem ferritin nanoparticle) and the seasonal flu vaccine Flucelvax.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years inclusive.
* Previous influenza immunization status:

  1. MN participants must have received at least 3 licensed seasonal flu vaccine doses over the past 5 years (fall or winter of 2021-2025).
  2. MN participants should have a gap of at least 6 months between their last seasonal flu vaccine and study enrollment.
  3. Uganda participants must have no prior exposure to any flu vaccine.
* The participant is able and willing to provide informed consent.
* Medical chart review and medical history without clinically significant findings or concerns.
* Physical examination without clinically significant findings or concerns.
* Body mass index (BMI) ≤ 30 kg/m2. This inclusion criterion can be voided if the participant is otherwise eligible and the study team finds the participant suitable for the LN biopsy via LN palpation on the physical exam.
* Screening laboratory results (blood) within institutional normal ranges (unless specified below otherwise). Screening lab tests include: CBCD, comprehensive metabolic panel (i.e., AST, ALT, ALP, BUN, creatinine, glucose, Na, K, Ca, total protein, albumin, total bilirubin), and HIV Ag/Ab test. Acceptance of screening lab results outside of the ranges below will need to be accompanied by a site investigator's approval.

  1. Hb ≥ 11 g/dL (males) or ≥ 10.5 g/dL (females).
  2. White blood cell (WBC) count in the range of 4,000-11,000 cells/μL.
  3. Normal WBC differential per institutional ranges.
  4. Total lymphocyte count ≥ 800 cells/μL.
  5. Platelet count in the range of 125,000-500,000 cells/μL.
  6. Na = 135-145 mmol/L
  7. K = 3.4-5.3 mmol/L
  8. Creatinine = 0.67-1.28 mg/dL
  9. Blood urea nitrogen (BUN) ≤ 20 mg/dL
  10. Glucose (non-fasting) = 65-116 mg/dL
  11. Ca = 8.6-10.0 mg/dL
  12. Total protein ≥ 6.0 g/dL
  13. Albumin ≥ 3.5 g/dL
  14. Total bilirubin ≤ 1.2 mg/dL
  15. ALP ≤ 165 U/L
  16. AST ≤ 50 U/L
  17. ALT ≤ 87 U/L
  18. Negative for HIV infection per study testing (FDA approved method of detection): non-reactive licensed 4th generation (Ag/Ab) HIV rapid test, EIA, or CIA.
* Women of reproductive potential / premenopausal:

  1. Negative beta-human chorionic gonadotropin (β-HCG) urine or serum pregnancy test at screening.
  2. Agrees to avoid pregnancy during the study.
  3. Agrees to use an effective means of birth control from at least 21 days prior to baseline visit through the end of the study (week 40). Acceptable birth control for this study is defined as:

     * Sexual abstinence with male partners.
     * Surgical sterilization (tubal ligation).
     * Male condom with or without a spermicidal agent.
     * Female condom.
     * Diaphragm or cervical cap.
     * Intrauterine device (IUD) (published data shows that expected failure rate is < 1% per year).
     * Hormone-based contraceptives including oral pills, injectables, implants, rings, and patches.
     * Partner has vasectomy.
* The participant is agreeable to the following study requirements:

  1. The participant should not receive an off-study flu vaccine until they complete the study (40 weeks from enrollment).
  2. The participant is available and willing to attend research visits for 40 weeks after enrollment and undergo all study procedures to provide samples, which are to be used for research-only purposes and can be stored indefinitely.
  3. The participant is able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
  4. The participant should not receive any other investigational research agents until they complete the study.
  5. The participant does not foresee becoming ineligible during study participation.

Exclusion Criteria:

* Breast-feeding or planning to become pregnant during the study.
* Any of the following substances are exclusionary if currently used or planned to be used at any time during the 40-week study period:

  1. Systemic immunosuppressive medications within the 4 weeks prior to enrollment (e.g., corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon, methotrexate, cancer chemotherapy). Use of inhaled, nasal spray, or topical steroids is not exclusionary.
  2. Any cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment.
  3. Blood products within 16 weeks prior to enrollment.
  4. Live attenuated vaccines within 4 weeks prior to enrollment.
  5. Inactivated vaccines within 2 weeks prior to enrollment.
  6. Investigational research agents within 4 weeks prior to enrollment.
  7. Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule.
  8. Current anti-tuberculosis prophylaxis or therapy.
  9. Previous investigational influenza vaccines.
  10. Previous investigational ferritin-based vaccines.
* History of any of the following clinically significant conditions:

  1. Severe allergic reactions to influenza vaccines in the past (e.g., Guillain-Barré syndrome, anaphylaxis, or angioedema)
  2. Other reactions to any vaccines that preclude receipt of the study vaccination as determined by the investigator.
  3. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
  4. Asthma that requires prednisone therapy 3 or more times in a 12-month period or rescue inhaler therapy more than weekly.
  5. Diabetes mellitus (type I or II), except for gestational diabetes.
  6. Thyroid disease that is not well controlled.
  7. Idiopathic urticaria within the past year.
  8. Autoimmune disease or immunodeficiency.
  9. Hypertension that is not well controlled (baseline systolic > 140 mmHg or diastolic > 90 mmHg).
  10. Bleeding disorder diagnosed by a healthcare professional (e.g., factor deficiency, coagulopathy, or platelet disorder) or significant bruising or bleeding difficulties with IM injections or blood draws.
  11. Active malignancy requiring systemic chemotherapy or surgery within preceding 12 months or expected during study participation. Minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) is permitted.
  12. Seizure disorder other than 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 12 months ago, or 3) seizures that have not required treatment within the last 12 months.
  13. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
  14. Guillain-Barré Syndrome.
  15. Current/active infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  16. Any medical, psychiatric, social condition, occupational reason, or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation, puts participant at risk, influences results of the study, or impairs a participant's ability to provide informed consent.
* History of ≥3 previous inguinal LN biopsies.
* Not a suitable surgical candidate per investigators' assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited local reactogenicity for 7 days after vaccine administration | Day 7
  Number of participants with solicited local symptoms per protocol
Occurrence of solicited systemic reactogenicity for 7 days after vaccine administration | Day 7
  Number of participants with solicited systemic symptoms per protocol
Occurrence of adverse events of all severities from baseline through 1-week follow-up after the 2nd LN biopsy on week 4 study visit | Week 5
  Number of participants with any adverse event through week 5
Occurrence of serious adverse events at any time throughout the study | Week 40
  Number of participants with any serious adverse event throughout the study

SECONDARY OUTCOMES:
Binding antibody responses to H1ssF at week 2 after vaccination in both cohorts (US and Uganda) | Week 2
  Antibody titer to H1ssF at week 2 after vaccination
Binding antibody responses to the Flucelvax HAs at week 2 after vaccination in both cohorts (US and Uganda) | Week 2
  Antibody titer to H1ssF at week 2 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tim Schacker, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No